CLINICAL TRIAL: NCT02684396
Title: A Phase 1, Randomized, Double-Blind, Placebo- Controlled, Safety, Tolerability, and Pharmacokinetic Study of Escalating Single Oral TAK-648 Doses in Healthy Subjects
Brief Title: Phase 1, TAK-648, Single-Rising Dose Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-648_101; U1111-1154-2329 (Other: WHO)
Record Dates: First submitted 2016-02-16; First posted 2016-02-18 (Estimated); Results first posted 2016-07-13 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-04

CONDITIONS: Healthy Volunteers
Keywords: Drug therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Cohort 1: TAK-648 0.05 mg (Experimental): TAK-648 0.05 mg, solution, orally, once on Day 1.
  Interventions: Drug: TAK-648
- Cohort 2: TAK-648 0.15 mg (Experimental): TAK-648 0.15 mg, solution, orally, once on Day 1.
  Interventions: Drug: TAK-648
- Cohort 3: TAK-648 0.35 mg (Experimental): TAK-648 0.35 mg, solution, orally, once on Day 1.
  Interventions: Drug: TAK-648
- Cohort 4: TAK-648 0.7 mg (Experimental): TAK-648 0.7 mg, solution, orally, once on Day 1.
  Interventions: Drug: TAK-648
- Cohort 5: TAK-648 0.85 mg (Experimental): TAK-648 0.85 mg, solution, orally, once on Day 1.
  Interventions: Drug: TAK-648
- Cohort 1-5: Placebo (Placebo Comparator): TAK-648 placebo-matching solution, orally, once on Day 1.
  Interventions: Drug: TAK-648 Placebo

INTERVENTIONS:
Drug: TAK-648 — TAK-648 Solution
  Arms: Cohort 1: TAK-648 0.05 mg; Cohort 2: TAK-648 0.15 mg; Cohort 3: TAK-648 0.35 mg; Cohort 4: TAK-648 0.7 mg; Cohort 5: TAK-648 0.85 mg
Drug: TAK-648 Placebo — TAK-648 placebo-matching solution
  Arms: Cohort 1-5: Placebo

SUMMARY:
The purpose of this study is to determine the safety, tolerability and pharmacokinetics of TAK-648 when administered as a single oral dose of TAK-648 solution at escalating dose levels in healthy participants.

DETAILED DESCRIPTION:
This was a phase 1, randomized, double-blind, placebo-controlled, single-center, single-dose study in healthy participants. The study is the first TAK-648 study in humans and is designed to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of a single dose of TAK-648 to healthy participants.

The compound being tested in this study is TAK-648. TAK-648 is being tested to find a safe and well-tolerated single dose.

This study measured how much of the study drug got into the blood stream and how long it took the body to get rid of it. Information about any side effects that may have occurred was also collected. This study was a randomized dose-rising study which means that the first group of research participants was assigned by chance to receive either the study drug or placebo. Placebo is a solution that looks like the study drug but has no active ingredient. The lowest dose of the study drug or placebo was given to the 1st group of participants (1st cohort) and a higher dose was given to the next group until all the doses of the study drug were tested. TAK-648 was dosed in 5 sequential cohorts with escalating doses from the lowest dose given in Cohort 1 to higher doses given in the subsequent cohort. Doses could be adjusted based on available safety, tolerability, and pharmacokinetic (PK) data.

Approximately 40 healthy male and female participants were planned for enrollment with 8 subjects planned (6 randomized to TAK-648 and 2 randomized to placebo) for each cohort. The study included 5 cohorts.

This single-center trial was conducted in the United States. The overall time to participate in this study was up to 45 days. Participants made multiple visits to the clinic, including one 5-day period of confinement to the clinic. All participants were contacted by telephone 14 days after the last dose of study drug and on Day 84 (+/-2 days) for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Is a healthy adult male or non-pregnant, non-lactating female.
2. Is aged 18 to 55 years, inclusive.
3. Weighs at least 55 kg (121 lbs) and has a body mass index (BMI) between 18.0 and 30.0 kg/m^2, inclusive.
4. Has a systolic blood pressure >90 and ≤150 mm Hg and a diastolic blood pressure of >60 and ≤90 mm Hg at Screening and at Check-in (Day -2).
5. Has a calculated creatinine clearance >60 mL/min at Screening and Check-in (Day -2).

Exclusion Criteria:

1. Has a known hypersensitivity to any component of the formulation of TAK-648, phosphodiesterase inhibitors or Listerine strips.
2. Has significant medical histories or currently uncontrolled clinical conditions, which may not be safe for participant to participate in the study, may impact the participant's ability to participate in the study; may influence absorption of the study drug, or may potentially confound the study results.
3. Has a history of persistent, chronic or intermittent nausea, vomiting, or diarrhea or had a current or recent (within 6 months) gastrointestinal disease that would influence the absorption of drugs
4. Has a diagnosis of major depression, bipolar disorder, or anxiety disorders or received any medication to treat any psychological disorders within 1 year prior to Screening.
5. Has abnormal laboratory values that suggest a clinically significant underlying disease or has the following laboratory abnormalities: alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) >2.5 times the upper limits of normal.
6. Use of any excluded medications, supplement, or food product outlined in the protocol.
7. Use of new medications during the course of the study including through the Follow-up period.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2014-08; Primary Completion 2015-04 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United States from 19 August 2014 to 08 July 2015.
Pre-assignment Details: Healthy Volunteers were enrolled in 1 of 6 treatment groups, once a day placebo, TAK-648 0.05 mg, 0.15 mg, 0.35 mg, 0.7 mg or 0.85 mg.
Period: Overall Study
Arm/Group | Cohort 1: TAK-648 0.05 mg | Cohort 2: TAK-648 0.15 mg | Cohort 3: TAK-648 0.35 mg | Cohort 4: TAK-648 0.7 mg | Cohort 5: TAK-648 0.85 mg | Cohort 1-5: Placebo
Started | 6 | 6 | 6 | 6 | 5 | 10
Completed | 6 | 6 | 6 | 6 | 5 | 10
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: TAK-648 0.05 mg | Cohort 2: TAK-648 0.15 mg | Cohort 3: TAK-648 0.35 mg | Cohort 4: TAK-648 0.7 mg | Cohort 5: TAK-648 0.85 mg | Cohort 1-5: Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 10 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.0 (13.21) | 32.5 (11.08) | 37.5 (9.07) | 37.0 (9.78) | 45.0 (11.51) | 36.2 (11.10) | 37.5 (10.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 4 | 2 | 2 | 11
  Male | 5 | 5 | 5 | 2 | 3 | 8 | 28
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 2 | 2 | 3 | 4 | 1 | 0 | 12
  Non-Hispanic and Latino | 4 | 4 | 3 | 2 | 4 | 10 | 27
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaskan Native | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 1 | 0 | 0 | 0 | 2 | 3
  Black or African American | 2 | 1 | 1 | 1 | 1 | 3 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 0 | 0 | 1
  White | 4 | 3 | 4 | 5 | 4 | 5 | 25
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 6 | 6 | 5 | 10 | 39
Height [Mean (Standard Deviation); unit: cm] | 177.2 (9.24) | 169.0 (8.58) | 172.2 (11.82) | 163.3 (8.21) | 170.6 (12.26) | 176.4 (8.46) | 172.0 (10.19)
Weight [Mean (Standard Deviation); unit: kg] | 76.1 (12.39) | 70.0 (9.32) | 75.6 (12.86) | 67.1 (4.36) | 76.1 (12.79) | 77.7 (14.33) | 74.1 (11.71)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 24.3 (3.60) | 24.5 (2.42) | 25.4 (2.37) | 25.3 (2.73) | 26.0 (2.26) | 24.8 (3.03) | 25.0 (2.69)
Hip Circumference [Mean (Standard Deviation); unit: cm] | 99.33 (6.683) | 96.33 (3.141) | 98.50 (8.385) | 102.83 (4.956) | 102.20 (4.207) | 98.63 (7.121) | 99.47 (6.180)
Waist Circumference [Mean (Standard Deviation); unit: cm] | 86.83 (9.174) | 82.50 (6.863) | 90.00 (5.762) | 86.17 (7.548) | 95.00 (3.391) | 88.06 (10.865) | 87.91 (8.420)
Waist to Hip Ratio [Mean (Standard Deviation); unit: ratio] | 0.87 (0.037) | 0.86 (0.061) | 0.92 (0.038) | 0.84 (0.074) | 0.93 (0.034) | 0.89 (0.069) | 0.88 (0.061)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Have at Least One Treatment-Emergent Adverse Event (TEAE)
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: Day 1 to Day 14
Population: Safety Analysis Set included all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: TAK-648 0.05 mg | Cohort 2: TAK-648 0.15 mg | Cohort 3: TAK-648 0.35 mg | Cohort 4: TAK-648 0.7 mg | Cohort 5: TAK-648 0.85 mg | Cohort 1-5: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 10
percentage of participants | 0 | 50.0 | 16.7 | 0 | 20.0 | 30.0

2. Primary Outcome: Percentage of Participants Who Meet the Markedly Abnormal Criteria, for Safety Laboratory Tests at Least Once Post-dose
Description: The percentage of participants with any markedly abnormal standard safety laboratory values (chemistry, hematology and urinalysis) collected throughout study.
Time Frame: Day 1 to Day 4
Population: Safety Analysis Set included all enrolled participants who received study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: TAK-648 0.05 mg | Cohort 2: TAK-648 0.15 mg | Cohort 3: TAK-648 0.35 mg | Cohort 4: TAK-648 0.7 mg | Cohort 5: TAK-648 0.85 mg | Cohort 1-5: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 10
percentage of participants
  Chemistry | 0 | 0 | 0 | 0 | 0 | 0
  Hematology | 0 | 16.7 | 0 | 0 | 0 | 0
  Urinalysis | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Percentage of Participants Who Meet the Markedly Abnormal Criteria for Vital Signs Measurements at Least Once Post-dose
Description: Vital signs will include body temperature (oral), sitting blood pressure (after the participant has rested for at least 5 minutes), respiration rate and pulse (bpm).
Time Frame: Day 1 to Day 4
Population: Safety Analysis Set included all enrolled participants who received study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: TAK-648 0.05 mg | Cohort 2: TAK-648 0.15 mg | Cohort 3: TAK-648 0.35 mg | Cohort 4: TAK-648 0.7 mg | Cohort 5: TAK-648 0.85 mg | Cohort 1-5: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 10
percentage of participants
  < Lower Criteria | 33.3 | 16.7 | 33.3 | 33.3 | 20.0 | 40.0
  > Upper Criteria | 0 | 0 | 0 | 0 | 40.0 | 20.0

4. Primary Outcome: Percentage of Participants With at Least One Occurrence of Severe Hypoglycemia Post-dose
Description: Severe hypoglycemia is defined as an event requiring assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions.
Time Frame: Day 1 to Day 4
Population: Safety Analysis Set included all enrolled participants who received study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: TAK-648 0.05 mg | Cohort 2: TAK-648 0.15 mg | Cohort 3: TAK-648 0.35 mg | Cohort 4: TAK-648 0.7 mg | Cohort 5: TAK-648 0.85 mg | Cohort 1-5: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 10
percentage of participants | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-648
Time Frame: Multiple time-points (up to 72 hours) post-dose
Population: PK Analysis Set included all enrolled participants who had at least 1 measureable plasma concentration.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1: TAK-648 0.05 mg | Cohort 2: TAK-648 0.15 mg | Cohort 3: TAK-648 0.35 mg | Cohort 4: TAK-648 0.7 mg | Cohort 5: TAK-648 0.85 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5
ng/mL | 0.619 (0.2461) | 2.330 (0.8022) | 3.997 (1.5958) | 11.845 (2.6415) | 11.712 (6.2166)

6. Secondary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-648
Time Frame: Multiple time-points (up to 72 hours) post-dose
Population: PK Analysis Set included all enrolled participants who had at least 1 measureable plasma concentration.
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1: TAK-648 0.05 mg | Cohort 2: TAK-648 0.15 mg | Cohort 3: TAK-648 0.35 mg | Cohort 4: TAK-648 0.7 mg | Cohort 5: TAK-648 0.85 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5
hours | 1.000 [0.50 to 2.00] | 1.500 [1.00 to 1.50] | 1.000 [0.50 to 1.50] | 1.000 [0.50 to 1.50] | 1.000 [1.00 to 1.50]

7. Secondary Outcome: AUClast: Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-648
Time Frame: Multiple time-points (up to 72 hours) post-dose
Population: PK Analysis Set included all enrolled participants who had at least 1 measureable plasma concentration.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Cohort 1: TAK-648 0.05 mg | Cohort 2: TAK-648 0.15 mg | Cohort 3: TAK-648 0.35 mg | Cohort 4: TAK-648 0.7 mg | Cohort 5: TAK-648 0.85 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5
ng*hr/mL | 4.452 (2.2891) | 16.614 (4.6927) | 27.927 (9.5790) | 75.280 (25.2406) | 92.661 (30.0958)

8. Secondary Outcome: AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-648
Time Frame: Multiple time-points (up to 72 hours) post-dose
Population: PK Analysis Set included all enrolled participants who had at least 1 measureable plasma concentration.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Cohort 1: TAK-648 0.05 mg | Cohort 2: TAK-648 0.15 mg | Cohort 3: TAK-648 0.35 mg | Cohort 4: TAK-648 0.7 mg | Cohort 5: TAK-648 0.85 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5
ng*hr/mL | 4.585 (2.2743) | 16.813 (4.6918) | 28.266 (9.5872) | 75.774 (25.3966) | 93.840 (30.8531)

ADVERSE EVENTS:
Time Frame: 14 Days
Description: At each visit the investigator had to document any occurrence of adverse events irrespective of the relation to study treatment.
Arm/Group | Cohort 1: TAK-648 0.05 mg | Cohort 2: TAK-648 0.15 mg | Cohort 3: TAK-648 0.35 mg | Cohort 4: TAK-648 0.7 mg | Cohort 5: TAK-648 0.85 mg | Cohort 1-5: Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/5 | 0/10
Other Adverse Events (participants affected / at risk) | 0/6 | 3/6 | 1/6 | 0/6 | 1/5 | 3/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: TAK-648 0.05 mg (N=6) | Cohort 2: TAK-648 0.15 mg (N=6) | Cohort 3: TAK-648 0.35 mg (N=6) | Cohort 4: TAK-648 0.7 mg (N=6) | Cohort 5: TAK-648 0.85 mg (N=5) | Cohort 1-5: Placebo (N=10)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Blood pressure orthostatic abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Blood pressure orthostatic decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.